CLINICAL TRIAL: NCT00170690
Title: Präferenz-Studie Bei älteren Patientinnen Mit Ovarialkarzinomrezidiv: Treosulfan Oral vs. intravenös
Brief Title: Preference Study With Elderly Patients Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: W. Lichtenegger, Prof. Dr., Charité-Universitätsmedizin Berlin, Augustenburger Platz 1, 13353 Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3401000
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Treosulfan 7000 mg/m² i.v. on day 1, 29, 57 etc
  Interventions: Drug: Treosulfan
- 2 (Experimental): Treosulfan 600 mg/m² p.o. on day 1-28, 57-84, etc
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — Treosulfan 600 mg/m² p.o. on daý 1-28, 57-84, etc
  Arms: 2
Drug: Treosulfan — Treosulfan 7000 mg/m² i.v. on day 1, 29, 57 etc
  Arms: 1

SUMMARY:
Comparison of the patient compliance treosulfan oral vs. intravenous (defined as end of therapy for the patient)

DETAILED DESCRIPTION:
Approximately 60% of all cancer diseases appear to people aged 65 years and older. Ovarian cancer is the most frequent cause of death among gynaecological malignant tumours. Since the highest carcinoma incidence is between the 60th and 70th year more women will come down with ovarian cancer because of increased life expectancy. At least 65% of patients with FIGO stage III/IV will exhibit a relapse or progress after first-line therapy. In most studies the age of the patients is limited to 65 years. It could be shown that especially elder patients often receive an inadequate operative and cytostatic therapy resulting in a worse prognosis.

Patients aged 70 years or elder who will be treated with treosulfan, given oral or intravenous, shall be compared regarding the patient compliance, toxicity especially hematological and gastrointestinal toxicity grade 3-4 (CTC NCI), overall survival, progression free survival, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patient with relapsed ovarian cancer
* study therapy of third regime
* measurable or evaluable tumor lesions or progression defined as CA-125 more than >= 100 U/ ml.
* Age >= 70 years
* ECOG 0-2
* written informed consent

Exclusion Criteria:

* Pretreatment with treosulfan
* patient without measurable or evaluable tumor lesions or CA-125 more than >= 100 U/ ml.
* no adequate bone marrow function (leukocyte <= 2,9 x 109/l, platelets <= 100 x 109/ l
* creatinin and bilirubin within >= 1,25 x fold of the reference laboratory´s normal range
* simultaneous radiotherapy

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2004-08; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Comparison of patient´s compliance in both arms defined as therapy break-offs | during study treatment

SECONDARY OUTCOMES:
Toxicity, overall survival, progression-free survival | during study treatment and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, Germany